CLINICAL TRIAL: NCT02964715
Title: The Effect of Empagliflozin on NAFLD in Asian Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Shireene Vethakkan, Associate Professor Dr., University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERF-4
Record Dates: First submitted 2016-10-30; First posted 2016-11-16 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Type2 Diabetes; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — empagliflozin

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional arm (Experimental): Patients with NAFLD and Type 2 Diabetes prescribed 25mg empagliflozin(JARDIANCE) daily for 6 months
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — 25 mg daily for 6 months
  Other Names: Jardiance

SUMMARY:
Non-Alcoholic Fatty Liver Disease( NAFLD) is common in patients with type 2 diabetes. Empagliflozin, an FDA-approved oral medication used to treat type 2 diabetes, has been shown to reduce production and deposition of fat in the liver in animal experiments. There is little published evidence that this is so in Asian patients with type 2 diabetes. The investigators designed this pilot study to determine if use of empagliflozin for 6 months in patients with type 2 diabetes can improve scan, blood marker and biopsy features of NAFLD.

DETAILED DESCRIPTION:
Empagliflozin, an FDA-approved SGLT2 (Sodium glucose transporter 2) inhibitor used to treat type 2 diabetes, has been shown to reduce hepatic de novo lipogenesis and hepatic steatosis in animal models. There is little published evidence that this is so in Asian patients with type 2 diabetes. The investigators designed this open label proof of concept trial to determine if use of empagliflozin for 6 months in patients with type 2 diabetes can improve biomarkers and histological features of biopsy proven NAFLD.

Hypotheses

1. 6 months of empagliflozin will result in improved histology on liver biopsy in type 2 dm patients with NAFLD

2.6 months of empagliflozin will result in changes in liver enzymes, adipocytokines and FGF levels in type 2 dm patients with NAFLD

3.6 months of empagliflozin will result in improved liver stiffness measurement in type 2 dm patients with NAFLD

Study protocol

This is a prospective open-label proof-of-concept study. The investigators plan to recruit 25 Asian patients with biopsy-proven NASH and type 2 diabetes and commence them on empagliflozin 25 mg daily for 6 months. Upon recruitment clinical information will be obtained via an interview and use of a structured questionnaire. Anthropometric measurements will be obtained at baseline and 6 months. A repeat liver biopsy will be performed after 6 months of empagliflozin therapy. MRI and fibroscan of the liver will be conducted at baseline and 6 months. Fasting blood samples will be drawn for glucose, insulin, c-peptide, triglyceride, HDL, LDL, total cholesterol, NEFA(non-esterified fatty acid), HbA1c , liver function test(including albumin, AST, ALT, gamma GT, uric acid, inflammatory markers, FGF(fibroblast growth factor) and other biomarkers at baseline and 6 months.

Patients will be reviewed by a physician at 1 month and 6 months for development of any potential adverse events while on empagliflozin therapy.

Patients will be instructed not to make any significant changes to diet and lifestyle in these 6 months in order to assess to full effect of the intervention with no possible confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven NASH
* Type 2 DM
* HbA1c :>6.5%
* BMI < 45kg/m2
* Any anti-diabetic agent except SGLT2 inhibitors, TZDs(thiazolidinediones), DPP4(Dipeptidyl peptidase4) inhibitors and GLP1 RAs(Glucagon-like Peptide 1-Receptor Agonists)

Exclusion Criteria:

* eGFR <45 ml/min
* structural and functional urogenital abnormalities, that predispose for urogenital infections
* Investigational product use in the last 6 months
* SGLT2 inhibitor, TZD, DPP4 inhibitor and GLP1 RA use within the past 6 months
* DKA(Diabetic Ketoacidosis) or HHS(Hyperosmoloar Hyperglycaemic Syndrome) within the last 6 months
* Pregnancy
* Presence of major contraindications to magnetic resonance imaging (cardiac pacemakers, claustrophobia, foreign bodies and implanted medical devices with ferromagnetic properties).
* Liver cirrhosis
* Type 1 diabetes
* Severe uncorrected insulin insufficiency
* Significant alcohol intake
* HIV infection
* Use of Traditional Chinese Medication or alternative therapies
* Coexisting causes of chronic liver disease - chronic viral hepatitis(B & C), autoimmune liver disease, hemochromatosis, Wilson's etc.
* Use of medications associated with steatosis eg. Methotrexate, anticonvulsants, antiretroviral therapy etc.
* h/o stroke
* Steroid therapy
* Endogenous Cushing's
* Familial hypertriglyceridemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in histological Grade as evaluated with Non-alcoholic Steatohepatitis Clinical Research Network Scoring System | baseline, 6 months
  liver biopsy
Change in serum FGF 21 | baseline and 6 months
  blood test

SECONDARY OUTCOMES:
Change in fibroscan and elastography measure of liver stiffness | baseline and 6 months
  imaging
Change in Liver enzymes | baseline and 6 months
  blood test - AST,ALT, gamma GT
Change in steatosis | baseline and 6 months
  histological
Change in lobular inflammation | baseline and 6 months
  histological
Change in ballooning | baseline and 6 months
  histological
Change in fibrosis | baseline and 6 months
  histological
Change in metabolic outcome -HbA1c | baseline and 6 months
  serum concentration
Change in metabolic outcome - fasting NEFA | baseline and 6 months
  serum concentration
Change in metabolic outcome - fasting Tg | baseline and 6 months
  serum concentration
Change in serum FGF 19 | baseline and 6 months
  serum concentration
Change in serum adiponectin | baseline and 6 months
  serum concentration
Change in serum IL-6 | baseline and 6 months
  serum concentration
Change in serum TNF alpha | baseline and 6 months
  serum concentration
Change in serum uric acid | baseline and 6 months
  serum concentration
Change in MRI features of NASH | baseline and 6 months
  serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Shireene R Vethakkan, MD, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940
- [Background] Ferrannini E, Mark M, Mayoux E. CV Protection in the EMPA-REG OUTCOME Trial: A "Thrifty Substrate" Hypothesis. Diabetes Care. 2016 Jul;39(7):1108-14. doi: 10.2337/dc16-0330. PMID 27289126
- [Background] Tahara A, Kurosaki E, Yokono M, Yamajuku D, Kihara R, Hayashizaki Y, Takasu T, Imamura M, Li Q, Tomiyama H, Kobayashi Y, Noda A, Sasamata M, Shibasaki M. Effects of SGLT2 selective inhibitor ipragliflozin on hyperglycemia, hyperlipidemia, hepatic steatosis, oxidative stress, inflammation, and obesity in type 2 diabetic mice. Eur J Pharmacol. 2013 Sep 5;715(1-3):246-55. doi: 10.1016/j.ejphar.2013.05.014. Epub 2013 May 23. PMID 23707905
- [Background] Hazlehurst JM, Woods C, Marjot T, Cobbold JF, Tomlinson JW. Non-alcoholic fatty liver disease and diabetes. Metabolism. 2016 Aug;65(8):1096-108. doi: 10.1016/j.metabol.2016.01.001. Epub 2016 Jan 11. PMID 26856933
- [Background] Ballestri S, Nascimbeni F, Romagnoli D, Lonardo A. The independent predictors of non-alcoholic steatohepatitis and its individual histological features.: Insulin resistance, serum uric acid, metabolic syndrome, alanine aminotransferase and serum total cholesterol are a clue to pathogenesis and candidate targets for treatment. Hepatol Res. 2016 Oct;46(11):1074-1087. doi: 10.1111/hepr.12656. Epub 2016 Mar 30. PMID 26785389
- [Background] Jojima T, Tomotsune T, Iijima T, Akimoto K, Suzuki K, Aso Y. Empagliflozin (an SGLT2 inhibitor), alone or in combination with linagliptin (a DPP-4 inhibitor), prevents steatohepatitis in a novel mouse model of non-alcoholic steatohepatitis and diabetes. Diabetol Metab Syndr. 2016 Jul 26;8:45. doi: 10.1186/s13098-016-0169-x. eCollection 2016. PMID 27462372
- [Background] Alisi A, Ceccarelli S, Panera N, Prono F, Petrini S, De Stefanis C, Pezzullo M, Tozzi A, Villani A, Bedogni G, Nobili V. Association between Serum Atypical Fibroblast Growth Factors 21 and 19 and Pediatric Nonalcoholic Fatty Liver Disease. PLoS One. 2013 Jun 26;8(6):e67160. doi: 10.1371/journal.pone.0067160. Print 2013. PMID 23840612
- [Background] Dushay JR, Toschi E, Mitten EK, Fisher FM, Herman MA, Maratos-Flier E. Fructose ingestion acutely stimulates circulating FGF21 levels in humans. Mol Metab. 2014 Oct 8;4(1):51-7. doi: 10.1016/j.molmet.2014.09.008. eCollection 2015 Jan. PMID 25685689
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Vanni E, Bugianesi E, Kotronen A, De Minicis S, Yki-Jarvinen H, Svegliati-Baroni G. From the metabolic syndrome to NAFLD or vice versa? Dig Liver Dis. 2010 May;42(5):320-30. doi: 10.1016/j.dld.2010.01.016. Epub 2010 Mar 6. PMID 20207596
- [Derived] Lai LL, Vethakkan SR, Nik Mustapha NR, Mahadeva S, Chan WK. Empagliflozin for the Treatment of Nonalcoholic Steatohepatitis in Patients with Type 2 Diabetes Mellitus. Dig Dis Sci. 2020 Feb;65(2):623-631. doi: 10.1007/s10620-019-5477-1. Epub 2019 Jan 25. PMID 30684076